CLINICAL TRIAL: NCT01403740
Title: Observational Acquired Haemophilia Registry
Brief Title: Turkish Acquired Haemophilia Registry
Acronym: EHEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Turkish Society of Hematology (Other)
Responsible Party: Turkish Society of Hematology, Turkish Society of Hematology
Other Study IDs: 2011/HEM/001
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-06

CONDITIONS: Acquired Haemophilia
Keywords: acquired haemophilia; factor VIII
MeSH Terms: conditions — Hemophilia A | interventions — Deamino Arginine Vasopressin; Azathioprine; Rituximab; Cyclosporine

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Blood sample for coagulation factor determination
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acquired haemophilia patients
  Interventions: Drug: rFVIIIa, aPCC, FVIII, DDAVP, Azathioprine, Rituximab, Cyclosporin

INTERVENTIONS:
Drug: rFVIIIa, aPCC, FVIII, DDAVP, Azathioprine, Rituximab, Cyclosporin — According to local clinical standards

SUMMARY:
Turkish Acquired Haemophilia Registry is a database in which information about clinical features and therapeutic management of acquired haemophilia is collected in Turkey.This is a multicentre, retrospective and prospective registry of subjects diagnosed and/or treated for acquired haemophilia. Patients will be registered and the response to different therapies, details of each bleeding episode and the outcome of haemostatic and immunosuppressive therapy (IST) will be recorded. Any male or female subject diagnosed with inhibitors to FVIII or other factors and treated for acquired haemophilia can be entered on the registry. Patients will be treated according to local practice. No additional tests or procedures are required by the registry. The retrospective period will not be time-limited and data will be collected from those recorded in the hospital notes. The prospective period will begin in September 1.2011, and will last for two years.

ELIGIBILITY:
Inclusion Criteria:

* Acquired haemophilia diagnosis, written consent

Exclusion Criteria:

* Being unable to give written consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acquired haemophilia diagnosed and/or treated in haematology clinics
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer A Demir, Prof, Principal Investigator — THD
Locations (1):
- Trakya University Haematology Clinic, Edirne, Turkey (Türkiye)